CLINICAL TRIAL: NCT04840043
Title: Assessment of Effectiveness of the Osteopathic Sympathetic Harmonization Applications on the Sympathetic Nervous System and the HPA Axis With Depression Diagnosed Adolescents: A Double-blind, Placebo-controlled, Randomized Study
Brief Title: Osteopathic Sympathetic Harmonization and Depression
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cumhuriyet University (Other)
Responsible Party: Principal Investigator, Ömer Osman PALA, Assistant Professor, Cumhuriyet University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: E-16-1106
Record Dates: First submitted 2021-04-04; First posted 2021-04-09 (Actual); Last update posted 2021-04-09 (Actual); Status verified 2021-04

CONDITIONS: Osteopathic Manipulative Treatment
Keywords: Depression; Sympathetic nervous system; Cortisol
MeSH Terms: conditions — Depression

STUDY DESIGN:
Intervention Model Description: A double-blind, placebo-controlled, randomized study
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double-blind trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Osteopathy Group (Experimental): Stimulation on the sympathetic truncus and prevertebral ganglia
  Interventions: Other: Osteopathic sympathic harmonization
- Control Group (Sham Comparator): Stimulation on similar areas with lighter touch and shorter duration
  Interventions: Other: Sham intervention

INTERVENTIONS:
Other: Osteopathic sympathic harmonization — Treatments that harmonize at the sympathetic nerves or plexus, e.g., sympathetic trunk stimulation by means of the rib-raise technique or stimulation of the prevertebral ganglia.
  Arms: Osteopathy Group
Other: Sham intervention — Different location, size and time of the rib-raise technique or stimulation of the prevertebral ganglia.
  Arms: Control Group

SUMMARY:
Depression appears to be resistant to the available pharmacological treatments. Autonomic responses accompanied by any psychological stress are sympathetic nervous system (SNS) and neuroendocrine responses are formed by hypothalamus-pituitary-adrenal (HPA) axis. The purpose of this study is; assessment of effectiveness of osteopathic approach on sympathetic nervous system and HPA axis in adolescents with depression.

DETAILED DESCRIPTION:
Depression diagnosed and volunteer to participate 39 cases who between the ages of 15-21 included. All participants were recruited and randomly assigned into two groups, the osteopathy group (OG) and the placebo group (PG). Stimulation on the sympathetic truncus and prevertebral ganglia were performed in the OG group. The stimulation of the PG group was performed with a lighter touch and a shorter duration in similar areas. Each participant was filled in the demographic data form, Beck Depression Scale and State and Trait Anxiety Inventory (STAI Form - 1 and Form - 2) before the application. Emotional state visual analog scale and STAI Form - 1 was filled and blood pressure and pulse measurement were made and saliva sample was taken before application, immediately after application and 20 minutes after application.

ELIGIBILITY:
Inclusion Criteria:

* To be diagnosed with clinical depression by a psychiatrist according to The Diagnostic and Statistical Manual of Mental Disorders (DSM-5) criteria
* Volunteering to participate in the study

Exclusion Criteria:

* Fever over 38.5
* Acute injury or infection
* Rib fracture
* Cardiac arrhythmia
* Using drugs that affect cortisol levels (oral contraceptives, hormonal drugs, antidepressants, antipsychotics etc.)
* Being pregnant, premenstrual or in the menstrual period for female participants

Ages: 15 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 39 (Actual)
Dates: Start 2017-10-11 (Actual); Primary Completion 2018-03-23 (Actual); Study Completion 2018-06-05 (Actual)

PRIMARY OUTCOMES:
The Beck Depression Inventory (BDI) | Before intervention
  The Beck Depression Inventory (BDI) is a 21-item, self-report rating inventory that measures characteristic attitudes and symptoms of depression.
The State-Trait Anxiety Inventory (STAI) Form - 1 | Before intervention
  The State-Trait Anxiety Inventory (STAI) is a commonly used measure of trait and state anxiety. It can be used in clinical settings to diagnose anxiety and to distinguish it from depressive syndromes. It also is often used in research as an indicator of caregiver distress.
Change from Baseline The State-Trait Anxiety Inventory (STAI) Form - 2 at 20 minutes | Before intervention, immediately after the intervention, 20 minutes after the intervention
  The State-Trait Anxiety Inventory (STAI) is a commonly used measure of trait and state anxiety. It can be used in clinical settings to diagnose anxiety and to distinguish it from depressive syndromes. It also is often used in research as an indicator of caregiver distress.
Change from Baseline Heart rate and blood pressure measurements at 20 minutes | Before intervention, immediately after the intervention, 20 minutes after the intervention
  Heart rate (beats per minute) and blood pressure (mm/Hg) were measured with automatic blood pressure monitor (the Microlife BP 3BT0-A). It is a clinically validated and 1-star automatic blood pressure monitor
Change from Baseline Salivary Biomarkers at 20 minutes | Before intervention, immediately after the intervention, 20 second after the intervention
  Salivary a-amylase and cortisol levels were measured for each sample. These biomarkers were analysed Enzyme-Linked Immunosorbent Assay.
Demographic data | Before intervention
  Sex; male or female
Demographic data | Before intervention
  Age; years
Demographic data | Before intervention
  Height (m); weight (kg); body mass index (kg/m2)

CONTACTS AND LOCATIONS:
Overall Officials: Omer Osman PALA, PhD, Study Director — Cumhuriyet University, Faculty of Health Sciences, Physiotherapy and Rehabilitation; Seyit CITAKER, Prof, Principal Investigator — Gazi University, Faculty of Health Sciences, Physiotherapy and Rehabilitation; Esra GUNEY, Assoc. Prof, Principal Investigator — Gazi University, Faculty of Medicine, Child and Adolescent Psychiatry; Aylin SEPICI DINCEL, Prof, Principal Investigator — Gazi University, Faculty of Medicine, Medical Biochemistry; Güner Melike GUVELI, MD, Principal Investigator — Gazi University, Faculty of Medicine, Child and Adolescent Psychiatry; Burak ARSLAN, MD, Principal Investigator — Gazi University, Faculty of Medicine, Medical Biochemistry
Locations (1):
- Sivas Cumhuriyet University, Sivas, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: CSR, Analytic Code
Time Frame: January 1, 2022

REFERENCES:
- [Background] Henderson AT, Fisher JF, Blair J, Shea C, Li TS, Bridges KG. Effects of rib raising on the autonomic nervous system: a pilot study using noninvasive biomarkers. J Am Osteopath Assoc. 2010 Jun;110(6):324-30. PMID 20606239
- [Derived] Pala OO, Citaker S, Guney E, Sepici A, Guveli GM, Arslan B, Guru M. Effectiveness of osteopathic manipulative applications on hypothalamic-pituitary-adrenal (HPA) axis in youth with major depressive disorder: a randomized double-blind, placebo-controlled trial. J Osteopath Med. 2024 Feb 29;124(6):267-275. doi: 10.1515/jom-2023-0056. eCollection 2024 Jun 1. PMID 38414339